CLINICAL TRIAL: NCT05270473
Title: Efficacy of Different Uterine Compression Sutures in Controlling Excessive Uterine Bleeding During Caesarean Section
Brief Title: Efficacy of Compression Sutures in Controlling Excessive Uterine Bleeding During Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Amany Salah El Din Abd El Hafeez Abd El Hady,MSC, MD Student, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD250/2019
Record Dates: First submitted 2021-10-08; First posted 2022-03-08 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Bleeding in Cesarean Section

STUDY DESIGN:
Intervention Model Description: randomised controlled trials 2 groups
Who Masked: Outcomes Assessor
Masking Description: Double blinding is difficult because the observer will see the type of procedure done. However, the measured outcomes are objective and unlikely to be biased by lack of blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A: b lynch (Active Comparator): B lynch uterine compressive suture was done
  Interventions: Procedure: uterine compressive sutures
- group B : Nusicaa suture (Active Comparator): Nusicaa uterine compressive suture was done
  Interventions: Procedure: uterine compressive sutures

INTERVENTIONS:
Procedure: uterine compressive sutures — uterine compression sutures comaprison
  Other Names: b lynch and nusicaa sutures

SUMMARY:
The investigators found that B- Lynch suture is more effective than Nausicca suture in controlling excessive uterine bleeding during cesarean section and avoiding the need of hysterectomy.

Also, the investigators found that B- lynch suture needs shorter procedure time with less blood loss compared to Nausicca suture.

Consequently the investigators recommend the use of B-Lynch suture as a compressive uterine suture to control excessive uterine bleeding during cesarean section and avoid the need of hysterectomy.

As a result of this study the investigators recommend further studies to compare different uterine compressive suture to verify the most effective uterine compressive suture.

DETAILED DESCRIPTION:
The objective of this study is to compare the efficacy of Nausicaa suture and B -lynch suture in controlling excessive uterine bleeding during cesarean section and avoiding the need for hystserctomy.

The investigators established this randomized controlled trial on participants with excessive uterine bleeding during cesarean section not responding to uterine massage and ecbolics in obstetric operative theatre in Ain Shams Maternity Hospitals.

During cesarean section, sixty participants who suffered from excessive uterine bleeding during cesarean section and not responding to uterine massage and ecbolics and who are willing to participate in the study and gave informed consent had Nausicaa or B-Lynch uterine compressive suture after randomizations using opaque sealed envelopes.

The selection of the type of suture done after allocation of women into two groups as llows:

Group (A):

Participants allocated in this group will have Nausicca suture done. Nausicaa suture will be applied by using round bodied, 3/8 circle curved needle, 70mm with 2-metric polyglactan suture. Suturing will be done by needle transfixing from the uterine serosa lateral to the bleeding area (or invaded myometrium) inside the uterine cavity. The needle will then be threaded along a horizontal course inside the uterine cavity until it encompassed the bleeding area, finally emerges at the other side of the uterine serosa. The sutures penetrated the full thickness of the myometrium without stitching the anterior and posterior walls together. Care will be taken to avoid transfixing any engorged parametrial vessels. A flat surgical knot will be then tied as tightly as possible above the serosa. Using these healthy myometrium as the anchoring points for needle transfixation, we will not encounter tissue destruction by the ligature. To achieve a better compression effect, the assistant often needed to clench the sutured myometrium while the operator ties off the knots. Additional sutures will made approximately 1.5-2 cm parallel to the previous stitches until haemostasis is achieved.

Group (B):

Participants allocated in this group will have B- lynch suture done. B-Lynch suture will be applied by using round bodied, 3/8 circle curved needle, 70mm with 2-metric polyglactan suture. Suturing will done according to method described by B-lynch et al. (1997) by starting in the uterus 3 cm from the right lower edge of the uterine incision and 3 cm from the right lateral border then passes through the uterine cavity to emerge at the upper incision margin 3 cm above and approximately 4 cm from the lateral border (because the uterus widens from below upwards), It will is be passed over to compress the uterine fundus, suture will pass posteriorly and vertically to enter the posterior wall of the uterine cavity at the same level as the upper anterior entry point, it will be pulled under moderate tension assisted by manual compression exerted by the first assistant. The suture will be passed through posteriorly and vertically over the fundus to lie anteriorly and vertically compressing the fundus on the left side as occurred on the right. The needle is passed in the same fashion on the left side through the uterine cavity and out approximately 3 cm anteriorly and below the lower incision margin on the left side. The two lengths of the suture are will be tight, assisted by bi-manual compression to minimise trauma and to achieve or aid compression and the principal surgeon will throw a surgical knot.

The two sutures were compare regarding need for hysterectomy, amount of blood loss will be assessed by number of soaked towels and suction titration, peripartum haemoglobin level drop (%) and haematocrit value change (%), number of received blood components (packed RBCs- fresh frozen plasma and platelets), procedure time (minutes), need for devascularisation, venous thromboembolism, postoperative pain and fever, hospital stay, number and cost of suture material used.

ELIGIBILITY:
Inclusion Criteria:

- Patients delivering by cesarean section with postpartum haemorrhage(intended for conservative management) as in

1. Non morbidly adherent placenta praevia.
2. Cases of uterine atony as in (Failed tocolysis, Twins, Polyhydramnios and History of postpartum haemorrhage).

After failed conservative management of excessive uterine massage and ecbolics

Exclusion Criteria:

* 1- Severely haemodynamic instablility needing immediate hysterectomy. 2- Morbidly adherent placenta: accrete, increta or percreta. 3- Patients with coagulopathy:
* Receiving anticoagulant therapy.
* With thrombocytopenia or thrombasthenia.
* known coagulation factor defect. 4 -Distorted uterus as unicornuate, bicornuate, fibroid uterus and adenomyosis uteri.

Ages: 16 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
need for hysterctomy | within 24 hours
  need for hysterctomy to control bleeding in cesarean section(YES/NO)

SECONDARY OUTCOMES:
blood loss | within 6 hours
  blood loss in ml
peripartum heamoglobin drop | within 6 hours
  differnce between pre and post operative heamoglobin (gm%)
procedure time | 1 hour
  timing of suture (minutes)
need for devascularisation | 1 hour
  need for devascularisation (YES/NO)
ICU admission | 24 hours
  need for ICU admission(YES/NO)
Venous thromboembolism | 6 weeks
  Venous thromboembolism (YES/NO)
postoperative fever | 48 hours
  temperature measurement in celsius

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed zeinhom, MD, Study Director — Ain Shams University
Locations (2):
- Egypt (2):
  - Dr Amany Salah, Cairo, Nasr City
  - Faculty of Medicine, Cairo

IPD SHARING:
Plan to Share IPD: Yes
yes to be publisged
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months